CLINICAL TRIAL: NCT05531721
Title: Retrospective Analysis of the Outcome of Patients Diagnosed With Hemophagocytic Lymphohistiocytosis (HLH) Treated at the S.C.Pediatric Oncohematology of the Regina Margherita Torino Hospital (OIRM)
Brief Title: HLH Patients - a Retrospective Study
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna (Other)
Responsible Party: Principal Investigator, Prof. Franca Fagioli, Clinical Professor, Azienda Ospedaliera Ospedale Infantile Regina Margherita Sant'Anna
Other Study IDs: HLH-OIRM
Record Dates: First submitted 2022-08-19; First posted 2022-09-08 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Hemophagocytic Lymphohistiocytoses
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- pediatric patients affected by hemophagocytic lymphohistiocytoses: pediatric patients with HLH
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation and retrospective data collection

SUMMARY:
Monocentric, observational, retrospective, no profit study aimed to analyze factors that are significantly impacting the outcome of patients diagnosed with HLH.

DETAILED DESCRIPTION:
retrospective data collection to study: type of HLH familial vs secondary, sex, age, presence of infectious cause, involvement central nervous system ( SNC), hepatic involvement, presence of hemophagocytosis, presence of splenomegaly, presence of involvement of other organs, the value of neutrophils (PMN), the value of hemoglobin, platelets, albumin, triglycerides, ferritin, LDH, type of therapy and the response to therapy after 2 months

ELIGIBILITY:
Inclusion Criteria:

* Have received HLH diagnosis according to HLH 2004 criteria
* age ⥶18 years.
* followed at our facility between January 2004 and December 2021
* Whose parents have consented to participation and data processing

Exclusion Criteria:

* The study does not foresee specific exclusion criteria other than the non-compliance with the inclusion criteria

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: pediatric patients with HLH
Sampling Method: Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2023-02-24 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
physiological parameter that are significantly impacting the outcome of patients diagnosed with HLH | through study completion, an average of 1 year
  Type of HLH (familial vs secondary); sex (M or F); age (in year); presence of infectious cause; involvement central nervous system (yes or no); hepatic involvement (yes or no); presence of hemophagocytosis (yes or no); presence of splenomegaly (yes or no); involvement of other organs (yes or no); value of neutrophils (PMN, in 10^9/L), hemoglobin (in g/dL), platelets (in 10^9/L), albumin (in g/L), triglycerides (in mg/dL), ferritin (in UI/L) and LDH (in UI/L);

CONTACTS AND LOCATIONS:
Overall Officials: Franca Fagioli, MD, Principal Investigator — AOU Città della Salute e della Scienza di Torino - OIRM
Locations (1):
- AOU Città della Salute e della Scienza di Torino - Presidio Infantile Regina Margherita, Turin, Italy

IPD SHARING:
Plan to Share IPD: No